CLINICAL TRIAL: NCT02323633
Title: A Single-blind, Randomised, Sham Controlled, Phase IIa Exploratory Clinical Trial, to Examine the Safety and Efficacy of BGX-3006 (tPCS) on Paediatric ADHD Participants.
Brief Title: Phase IIa Exploratory Clinical Trial, to Examine the Safety and Efficacy of tPCS on Paediatric ADHD Participants
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Braingear Technologies GmbH (Industry)
Collaborators: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BGX-3006
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Pediatric Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tPCS group (Active Comparator): Arm in which random noise oscillating frequencies will be produced for the duration of 20 minutes.
  Interventions: Device: Braingear Brainbuds Pulsed Current stimulation device
- Sham group (Sham Comparator): Arm in which no random noise oscillating frequencies will be produced for the duration of 20 minutes
  Interventions: Device: Sham

INTERVENTIONS:
Device: Braingear Brainbuds Pulsed Current stimulation device — Transcranial Pulsed Current stimulation (tPCS) at random noise oscillating frequencies for a duration of 20 minutues
  Arms: tPCS group
Device: Sham — No transcranial Pulsed Current Stimulation (tPCS)
  Other Names: Braingear Brainbuds Pulsed Current stimulation device
  Arms: Sham group

SUMMARY:
Children with ADHD display a certain brainwave profile which might be different to that of a child who does not have ADHD. Treatment with tPCS (transcranial pulsed current stimulation) has shown that this brainwave profile could possibly be altered to more closely resemble a brainwave profile of a child who does not have ADHD. Researchers believe that by changing this brainwave profile it might lessen symptoms of ADHD.

tPCS is a name used to describe the type of current this device produces. It involves randomly (in no specific pattern) produced pulses of current at different times that the brain picks up. These pulses of low current stimulate the brain in a certain way and affect the brainwave activity.

Treatment is given by applying a low frequency current using small electrodes clipped to the earlobes. The current comes from an external battery source. The pulses of current generated by this device stimulate certain parts of the brain which result in a possible increased control of attention and behaviour. This treatment has already been proven to be safe and will not hurt your child.

Due to these specific parts of the brain being stimulated, and the positive results of previous research, it seems possible to control certain functions in children suffering from inattention and hyperactivity.

The idea of using tPCS stimulation as a possible way for helping children with confirmed ADHD opens a new window to future research. The final goal of this device and research is to offer a safe, non-invasive (conservative treatment that does not require piercing into the body or the removal of tissue) treatment that can be used on a long-term basis and shows a clear improvement of ADHD symptoms for children and even adults with ADHD.

DETAILED DESCRIPTION:
- Inspection of Records: Investigators and institutions involved in the trial will permit trial-related monitoring, audits, Independent Ethics Committee (IEC) review, and regulatory inspection(s) by providing direct access to all trial records. In the event of an audit, the investigator agrees to allow the sponsor, representatives of the sponsor and applicable regulatory authorities access to all trial records. The confidentiality of records that can identify participants will be protected, respecting the privacy and confidentiality rules in accordance with regulatory requirements.

The investigator must promptly notify the sponsor of any audits scheduled by any regulatory authorities and promptly forward copies of any audit reports received to the sponsor.

In order to ensure data accuracy, data for individual participant visits must be completed as soon as possible/ during/ immediately following the visit. All completed data will be reviewed, signed, and dated by the investigator in a timely manner.

- Database Management and Quality Control: Data management, including the development and management of a database, will be performed in accordance with regulatory requirements. The designated data management vendor will review the CRF data for completeness and accuracy. A formal querying process will be followed whereby the data management group will request the site personnel to clarify any apparent erroneous entries or inconsistencies and will request additional information from the site as required.

Medical history/current medical conditions and adverse events will be coded using the Medical dictionary for regulatory activities (MedDRA) terminology.

- Sample Size: As this research is exploratory in nature a sample size was calculated based on some assumptions as there is no current data to compare in pediatrics, tPCS, and ADHD. Since no preliminary data is available a clinically relevant improvement is regarded as a 15% shift on the total range of the two ADHD sub-scales (Inattention and Hyperactivity/Impulsivity), with 9 items in each, i.e. 4.05 (=0.15 x 27 where items score 0 to 3 Likert scale). The standard deviation is estimated as range/6 = 27/6 = 4.5, i.e. the total range of a Gaussian distribution was 6 standard deviation. A sampling ratio of 2:1 is used. A sample size of 48 children (32:16) will have 80% power to detect a difference of 4.05 points between the groups when testing two-sided using Students t-test at the 0.05 level of significance.

Continuous data will be summarised using descriptive statistics. Categorical data will be presented using N and % (using the number of participants without missing data in the calculation). 95% confidence intervals will be determined for all data, where applicable. No imputation of missing values will be performed in the calculation of summary statistics.

- Safety Data Analysis: The safety analyses will be performed for the safety population only. All safety parameters (adverse events, physical examination findings, vital signs, physical measurements and qEEG findings) will be summarised descriptively by treatment group. The descriptive statistics will include the number of observations, mean, standard deviation, median, minimum and maximum for continuous variables and number of observations and their percentages for categorical variables. Changes from baseline as well as shift tables will be provided for the safety laboratory parameters (within, below or above normal range).

The analysis of adverse events will include all treatment emergent adverse events. Adverse events will be coded using MedDRA and will be presented by system organ class and preferred term for each treatment group.

- Efficacy Data

1. Primary Efficacy analysis:

   The mean change in both the Inattention and Hyperactivity-Impulsive subscales of the SNAP-IV-C rating scale as well as the Conners'3 Parent rating scale from baseline to Day 42 will be calculated for each group. Mean changes from baseline at the other trial time points (Days 0, 14, 28, and 42) will also be calculated.

   The statistical analysis methods will consist of paired t-tests within groups and analysis of Co-variance (ANCOVA) between groups for the change in assessments over time. The paired t-tests will compare the change variable from before tPCS administration to after tPCS within groups (active and sham condition). A one-way ANCOVA, with factor groups (active or sham) and co-variance baseline value, will be employed to compare groups with respect to change from baseline for estimated outcomes, e.g. change in complete scores from baseline to 6-weeks for inattentive and hyperactivity-impulsivity on SNAP-IV-C and Conners'3 Parent rating scales. Groups will also be compared over time (Days 0, 14, 28 and 42) using a linear mixed model analysis and of particular interest will be the interaction between group and time.
2. Secondary Efficacy analysis:

The mean change in the psychometric test-battery from baseline to Day 42 will be calculated for each group. Mean changes from baseline at the other trial time points (Days 0, 14, 28, and 42) will also be calculated.

The statistical analysis methods will consist of paired t-tests within groups and analysis of Co-variance (ANCOVA) between groups for the change in assessments over time. The paired t-tests will compare the change variable from before tPCS administration to after tPCS within groups (active and sham condition). A one-way ANCOVA, with factor groups (active or sham) and co-variance baseline value, will be employed to compare groups with respect to change from baseline for estimated outcomes, e.g. change in complete scores from baseline to 6-weeks for the psychometric test-battery. Groups will also be compared over time (Days 0, 14, 28 and 42) using a linear mixed model analysis for repeated measures and of particular interest will be the interaction between group and time.

EEG analysis Power spectra will be determined for each epoch of data for the frequency-domain analysis. Mean and median power frequencies will be calculated within each of the 4 EEG frequency bands (intraband) and over the entire EEG range (interband). Also, the band power fractions or relative amount of power within an EEG band with respect to the total amount of spectrum power will be determined. The coherence analysis will be completed using two bands (alpha and theta) and four sub-bands (low-alpha (8-10 Hz), high-alpha (10-12 Hz), low-beta (12-20 Hz), and high-beta (20-30 Hz)). We will use the Welch's averaged modified periodogram method to find the estimated coherence of signal x and y, representing each electrode site. It is a function of the power spectral densities of x and y and their cross power spectral density. Groups will also be compared over time (Days 0, 42 and 84) using a linear mixed model analysis for repeated measures and of particular interest will be the interaction between group and time.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the written informed consent process for trial participation, by parent(s) or legal guardian(s), prior to all trial-related procedures
* Completion of written assent for trial participation, by participant, prior to all trial-related procedures
* Male or female participants aged 6 to 12 years
* Newly diagnosed (Diagnosis made by DSM-V criteria), treatment naïve participants
* Participants and parent(s) or legal guardian(s) must have the ability to communicate well with the investigator and to understand and comply with the requirements of the trial
* Participants and parent(s) or legal guardian(s) must agree to stay in contact with the trial site for the duration of the trial and provide updated contact information as necessary.

Exclusion Criteria:

* Existence of a major neurologic or psychiatric condition (epilepsy, severe depression etc.)
* History of head injury resulting in more than a momentary loss of consciousness
* Previous neurosurgery
* Presence of unstable medical conditions, such as: Diabetes Mellitus, Cardiac Pathology, Cancer, Kidney Insufficiency, Acute Thrombosis
* Presence of any implanted metal or electronic medical devices present in the head, excluding any dental implants
* Subjects on any prohibited concomitant medication
* Any other medical condition which, in the opinion of the Investigator, could affect the participant's health during trial participation or could compromise his/her ability to participate in the trial
* In the opinion of the investigator, the participant and his/her parent(s) or legal guardian(s) is not reliable for participation in the trial

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy objective will be measured by the change in scores from baseline to Day 42 in both the SNAP-IV-C and Connors'3 Parent Rating Scales | 42 days
Safety and tolerability will be measured by the incidence and severity of adverse events and changes in physical examination findings, vital signs and qEEG findings. | 42 days

SECONDARY OUTCOMES:
The secondary efficacy objective will be measured by the change in scores from baseline to day 42 in the psychometric analysis conducted by the psychometrist | 42 days
The change from baseline to day 42 in the electrophysiological observations of a qEEG. | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Johan A Erasmus, MBChB, Principal Investigator — Netcare Moot Hospital

REFERENCES:
- [Background] Aosaki T, Graybiel AM, Kimura M. Effect of the nigrostriatal dopamine system on acquired neural responses in the striatum of behaving monkeys. Science. 1994 Jul 15;265(5170):412-5. doi: 10.1126/science.8023166.
- [Background] Zaghi S, Acar M, Hultgren B, Boggio PS, Fregni F. Noninvasive brain stimulation with low-intensity electrical currents: putative mechanisms of action for direct and alternating current stimulation. Neuroscientist. 2010 Jun;16(3):285-307. doi: 10.1177/1073858409336227. Epub 2009 Dec 29. PMID 20040569
- [Background] Wilens T, Pelham W, Stein M, Conners CK, Abikoff H, Atkins M, August G, Greenhill L, McBurnett K, Palumbo D, Swanson J, Wolraich M. ADHD treatment with once-daily OROS methylphenidate: interim 12-month results from a long-term open-label study. J Am Acad Child Adolesc Psychiatry. 2003 Apr;42(4):424-33. doi: 10.1097/01.CHI.0000046814.95464.7D. PMID 12649629
- [Background] Stergiakouli E, Thapar A. Fitting the pieces together: current research on the genetic basis of attention-deficit/hyperactivity disorder (ADHD). Neuropsychiatr Dis Treat. 2010 Sep 7;6:551-60. doi: 10.2147/NDT.S11322. PMID 20856918
- [Background] Sprich S, Biederman J, Crawford MH, Mundy E, Faraone SV. Adoptive and biological families of children and adolescents with ADHD. J Am Acad Child Adolesc Psychiatry. 2000 Nov;39(11):1432-7. doi: 10.1097/00004583-200011000-00018. PMID 11068899
- [Background] Shealy YF. Synthesis and evaluation of some new retinoids for cancer chemoprevention. Prev Med. 1989 Sep;18(5):624-45. doi: 10.1016/0091-7435(89)90034-0. PMID 2694159
- [Background] Voeller KK. Attention-deficit hyperactivity disorder (ADHD). J Child Neurol. 2004 Oct;19(10):798-814. doi: 10.1177/08830738040190100901. PMID 15559895
- [Background] Goodman R, Stevenson J. A twin study of hyperactivity--II. The aetiological role of genes, family relationships and perinatal adversity. J Child Psychol Psychiatry. 1989 Sep;30(5):691-709. doi: 10.1111/j.1469-7610.1989.tb00782.x. PMID 2793957
- [Background] Polania R, Nitsche MA, Korman C, Batsikadze G, Paulus W. The importance of timing in segregated theta phase-coupling for cognitive performance. Curr Biol. 2012 Jul 24;22(14):1314-8. doi: 10.1016/j.cub.2012.05.021. Epub 2012 Jun 7. PMID 22683259
- [Background] Loe IM, Feldman HM. Academic and educational outcomes of children with ADHD. J Pediatr Psychol. 2007 Jul;32(6):643-54. doi: 10.1093/jpepsy/jsl054. Epub 2007 Jun 14. PMID 17569716
- [Background] Biederman J, Spencer T. Attention-deficit/hyperactivity disorder (ADHD) as a noradrenergic disorder. Biol Psychiatry. 1999 Nov 1;46(9):1234-42. doi: 10.1016/s0006-3223(99)00192-4. PMID 10560028
- [Background] Brook U, Boaz M. Adolescents with attention deficit and hyperactivity disorder/learning disability and their proneness to accidents. Indian J Pediatr. 2006 Apr;73(4):299-303. doi: 10.1007/BF02825823. PMID 16816490
- [Background] Datta A, Dmochowski JP, Guleyupoglu B, Bikson M, Fregni F. Cranial electrotherapy stimulation and transcranial pulsed current stimulation: a computer based high-resolution modeling study. Neuroimage. 2013 Jan 15;65:280-7. doi: 10.1016/j.neuroimage.2012.09.062. Epub 2012 Oct 5. PMID 23041337
- [Background] Edelmuth RC, Nitsche MA, Battistella L, Fregni F. Why do some promising brain-stimulation devices fail the next steps of clinical development? Expert Rev Med Devices. 2010 Jan;7(1):67-97. doi: 10.1586/erd.09.64. PMID 20021241
- [Background] Arnsten AF, Steere JC, Hunt RD. The contribution of alpha 2-noradrenergic mechanisms of prefrontal cortical cognitive function. Potential significance for attention-deficit hyperactivity disorder. Arch Gen Psychiatry. 1996 May;53(5):448-55. doi: 10.1001/archpsyc.1996.01830050084013. PMID 8624188
- [Background] Arnsten AF, Li BM. Neurobiology of executive functions: catecholamine influences on prefrontal cortical functions. Biol Psychiatry. 2005 Jun 1;57(11):1377-84. doi: 10.1016/j.biopsych.2004.08.019. PMID 15950011
- [Background] Bader A, Adesman A. Complementary and alternative therapies for children and adolescents with ADHD. Curr Opin Pediatr. 2012 Dec;24(6):760-9. doi: 10.1097/MOP.0b013e32835a1a5f. PMID 23111680
- [Background] Ahuja A, Martin J, Langley K, Thapar A. Intellectual disability in children with attention deficit hyperactivity disorder. J Pediatr. 2013 Sep;163(3):890-5.e1. doi: 10.1016/j.jpeds.2013.02.043. Epub 2013 Apr 19. PMID 23608559
- [Background] Kessler RC, Adler L, Barkley R, Biederman J, Conners CK, Demler O, Faraone SV, Greenhill LL, Howes MJ, Secnik K, Spencer T, Ustun TB, Walters EE, Zaslavsky AM. The prevalence and correlates of adult ADHD in the United States: results from the National Comorbidity Survey Replication. Am J Psychiatry. 2006 Apr;163(4):716-23. doi: 10.1176/ajp.2006.163.4.716. PMID 16585449